CLINICAL TRIAL: NCT04438122
Title: Effect of Light to Moderate Wine Consumption on Cardiovascular Markers in Coronary Heart Disease Patients
Brief Title: Effect of Wine Consumption on Cardiovascular Markers in CHDs Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Elizabeth Fragopoulou, Assistant Professor of Biological Chemistry, Harokopio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HarokopioU
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Cardiovascular Disease
Keywords: wine; cardiovascular disease; inflammatory biomarkers; platelet aggregation; Platelet Activating Factor; ethanol; PBMCs; Wine microcontsituents
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Red Wine group (Active Comparator): Participants of this group consumed 200ml of red wine along with a meal (lunch or dinner) every day for 8 weeks.
  Interventions: Other: Cabernet Sauvignon
- Ethanol group (Active Comparator): Participants of this group consumed 69mL of tsipouro along with a meal (lunch or dinner) every day for 8 weeks.
  Interventions: Other: Tsipouro
- Control group (No Intervention): Participants of this group consumed no alcohol along with a meal (lunch or dinner) every day for 8 weeks

INTERVENTIONS:
Other: Cabernet Sauvignon — Cabernet Sauvignon is a red wine from a greek company which contains 13.5% alcohol vol.
  Arms: Red Wine group
Other: Tsipouro — Tsipouro is a greek spirit which contains 38% alcohol vol
  Arms: Ethanol group

SUMMARY:
Many epidemiological studies support that 20-30gr of alcohol consumption per day is related with lower risk for cardiovascular diseases, heart attack as well as mortality related to these diseases. Since the French paradox was reported, a number of experimental and clinical studies have demonstrated the protective effect of red wine compared to other alcoholic drinks on different pathways of the pathogenesis of atherosclerosis. The investigator's previous results revealed that wine contain micro-constituents that exert potent in vitro anti-platelet and anti-inflammatory actions. Also, the wine consumption along with a standardized meal reduced platelet aggregation and biosynthesis of Platelet Activating Factor in healthy men.

Although a large number of studies have reported protective effect of wine against atherosclerosis in healthy people there are few data about the effect of long-term moderate wine consumption in population with CVD. Therefore, the aim of this randomized, intervention clinical study, with control group was to report the effects of regular light to moderate wine consumption on cardiovascular biomarkers in people with CVD.

DETAILED DESCRIPTION:
The study was a randomized, controlled, three-arm parallel intervention study, designed to evaluate if the light to moderate wine consumption could modulate thrombosis and inflammation, in patients with cardiovascular disease. The study was carried out in accordance with the guidelines laid down in the Declaration of Helsinki (1989) of the World Medical Association and was approved by the Bioethics Committee of Harokopio University. Seventy one men patients with cardiovascular disease were initially recruited to participate in the study. The recruitment took place in several hospitals of Athens in Greece under the supervisor of corresponding cardiologist. Finally 64 met the inclusion criteria. Prior to intervention all participants signed an informed consent All volunteers followed an initial 15 days wash-out period, abstaining from alcohol; then, they randomly assigned to one of the three intervention groups. The randomization code was prepared by a staff member who was not involved in running the trial, by using computer-generated random numbers. Subjects instructed to follow their usual diet and not change their medication during the study. In Group A (control group), participants consumed no alcohol, in Group B (ethanol group) participants consumed 69 mL of tsipouro with 38% alcohol and participants in Group C consumed 200ml of red wine (Cabernet Sauvignon 13.5% alcohol vol.). The ethanol that was consumed in the last two groups was equal at 27gr of ethanol per day and alcoholic beverage was consumed along with the meal (lunch or dinner). Finally, 57 participants completed the study, in particular 20 in Group A, 16 in Group B and 21 in Group C. Intervention lasted two months and biological samples (blood, urine) were collected at the beginning (0 week), in the middle (4 week) and in the end (8 week) of each intervention.

ELIGIBILITY:
Inclusion Criteria:

The presence of Coronary Heart disease established by angiography or the presence of one of the following:

1. positive stress test
2. positive myocardial perfusion scintigraphy with Thallium
3. positive triplex heart ultrasound with Dobutamine

If nothing of the criteria above existed then hospitalization because of myocardial infarction or stroke.

Stable medication for at least 6 months.

Habit to drink 10-28gr of alcohol per week.

Exclusion Criteria:

History of any other inflammatory disease, diabetes, presence of cold or flu, acute respiratory infection, dental problems and renal/hepatic diseases.

Ages: 37 Years to 82 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Effect on platelet aggregation against PAF | Changes between baseline, 4 and 8 weeks.
  % Change of EC50 value of platelet aggregation against PAF
Effect on platelet aggregation against ADP | Changes between baseline, 4 and 8 weeks.
  % Change of EC50 value of platelet aggregation against ADP
Effect on platelet aggregation against collagen | Changes between baseline, 4 and 8 weeks.
  % Change of EC50 value of platelet aggregation against collagen
Effect on inflammatory markers (activity of Lyso-PAF-AT) | Changes between baseline, 4 and 8 weeks.
  % Change in the activity of PAF biosynthetic enzyme Lyso-PAF AT
Effect on inflammatory markers (activity of PAF-CPT) | Changes between baseline, 4 and 8 weeks.
  % Change in the activity of PAF biosynthetic enzyme PAF-CPT
Effect on inflammatory markers (activity of PAF-AH) | Changes between baseline, 4 and 8 weeks.
  % Change in the activity of PAF degradation enzyme PAF-AH
Effect on inflammatory markers (activity of LpPLA2) | Changes between baseline, 4 and 8 weeks.
  % Change in the activity of PAF degradation enzyme Lp-PLA2
Effect on inflammatory markers | Changes between baseline, 4 and 8 weeks.
  % Changes of Adiponectin, IL-6, CRP
Cytokine secretion by PBMC | Changes between baseline, 4 and 8 weeks.
  Secretion of TNFa and IL-1β by PBMC under basal and inflammatory (LPS-induced) conditions at 4 and 24h incubation
Effect on endothelial function markers | Changes between baseline, 4 and 8 weeks.
  % Changes of VCAM, P-selectin.

SECONDARY OUTCOMES:
Effect on biochemical indices | Changes between baseline, 4 and 8 weeks.
  % Changes of Total cholesterol, LDL-chol, HDL-chol, triacylglycerols, uric acid, glucose, insulin, SGOT/AST, SGPT/ALT, γ-GT
Effect on oxidative stress markers | Changes between baseline, 4 and 8 weeks.
  % Changes of TBARS, Lag time, GPx

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition-Dietetics, Harokopio University, Athens, Greece

IPD SHARING:
Plan to Share IPD: No